CLINICAL TRIAL: NCT05496738
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED, DOSE-ESCALATING STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF SINGLE AND MULTIPLE INTRAVENOUS AND SUBCUTANEOUS DOSES OF PF-07264660 IN HEALTHY PARTICIPANTS
Brief Title: A Preliminary Study to Evaluate PF-07264660 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: C4521001
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: Healthy volunteers; Inteurleukin-33; Inteurleukin-4; Inteurleukin-13; IL-33; IL-4; IL-13; monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Investigators and other site staff will be blinded to participants' assigned study intervention.
  Participants will be assigned to receive study intervention according to the assigned treatment group from the randomization scheme. Investigators will remain blinded to each participant's assigned study intervention throughout the course of the study.
  In the event of a Quality Assurance audit, the auditor(s) will be allowed access to unblinded study intervention records at the site(s) to verify that randomization/dispensing has been done accurately.
  Sponsor staff not directly involved in the conduct of the study will be unblinded to participants' assigned study intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- PF-07264660 intravenous single ascending dose (Experimental): PF-07264660 will be administered intravenously
  Interventions: Drug: PF-07264660 intravenous single ascending dose
- PF-07264660 subcutaneous multiple ascending dose (Experimental): PF-07264660 will be administered subcutaneously
  Interventions: Drug: PF-07264660 subcutaneous multiple ascending dose
- Intravenous placebo (Placebo Comparator): Placebo will be administered intravenously
  Interventions: Other: Intravenous placebo
- Subcutaneous Placebo (Placebo Comparator): Placebo will be administered subcutaneously
  Interventions: Other: subcutaneous placebo

INTERVENTIONS:
Drug: PF-07264660 intravenous single ascending dose — PF-07264660 will be administered intravenously in single ascending doses
  Arms: PF-07264660 intravenous single ascending dose
Drug: PF-07264660 subcutaneous multiple ascending dose — PF-07264660 will be administered subcutaneously in multiple ascending doses
  Arms: PF-07264660 subcutaneous multiple ascending dose
Other: Intravenous placebo — Placebo will be administered intravenously in single ascending doses
  Arms: Intravenous placebo
Other: subcutaneous placebo — Placebo will be administered subcutaneously in multiple ascending doses
  Arms: Subcutaneous Placebo

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of study medicine PF-07264660 compared to a placebo. This is the first study of PF-07264660 in humans. All participants in this study will received PF-07264660 or a placebo and it will be assigned by chance. People may be able to participate if they are healthy. The study medicine may be given by shots under the skin or through a vein depending on which group you are assigned to. If you are assigned into Part A, you will receive the study medicine once, stay overnight at the research unit from 3 to 5 overnight stays and you will need to visit the clinic about 11 follow-up visits. Participants will be in this study for up to about 541 days. If you are assigned into Part B, you will receive the study medicine three times, stay overnight at the clinic from 3 to 5 overnight stays and you will need to visit the research unit about 12 follow-up visits. Participants willbe in this study for up to about 561 days.

DETAILED DESCRIPTION:
This is an first-in-human within-cohort randomized, participant- and investigator-blind, sponsor-open, placebo-controlled study of the safety, tolerability, pharmacokinetics, and pharmacodynamics following single ascending dose and multiple ascending dose.

PF-07264660 that will be conducted in healthy adults. Up to approximately 67 participants will be enrolled into the study and randomly assigned to receive PF-07264660 or placebo. This will include up to approximately 43 healthy participants (including 5 optional Japanese participants) in Part A, and up to approximately 24 healthy participants (including 8 participants in optional multiple ascending dose cohort) in Part B.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer male and female participants between 18 to 65 years of age
* Body Mass Index (BMI) of 17.5 to 32 kg/m2; and a total body weight >50 kg (110 lb)

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Evidence of active, latent, or inadequately treated infection with Mycobacterium tuberculosis
* Participants with acute or chronic infections or infection history
* History of human immunodeficiency virus (HIV); Infection with hepatitis B or hepatitis C viruses according to protocol specific testing algorithm
* History of febrile illness within 5 days prior to the first dose of investigational product.
* Recent exposure to live or attenuated vaccines within 28 days of the screening visit.
* Failure to comply with coronavirus disease 2019 (COVID-19) vaccination requirements as per site protocols.
* Have any malignancies or have a history of malignancies with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin, or cervical carcinoma in situ.
* History of any lymphoproliferative disorder such as Epstein-Barr Virus (EBV) related lymphoproliferative disorder, history of lymphoma, leukemia, or signs and symptoms suggestive of current lymphatic or lymphoid tissue disease.
* Undergone significant trauma or major surgery within 1 month of the first dose of study drug
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer)
* Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≥1.5 × Upper limit of normal (ULN);
* Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ULN.
* estimated glomerular filtration rate (eGFR) ≤75 mL/min/1.73 m2 based on chronic kidney disease epidemiology (CKD-EPI) equation
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening
* Participants with more than 5 cigarettes per day or ≥10 pack years
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent treatment related adverse events (AE's) | Baseline up to approximately 1.5 years
  To evaluate the safety and tolerability of PF 07264660, following single and multiple doses in healthy adults
Number of participants with treatment emergent treatment-related serious adverse events (SAE's) | Baseline up to approximately 1.5 years
  To evaluate the safety and tolerability of PF 07264660, following single and multiple doses in healthy adults
Number of participants with change from baseline in blood pressure | Baseline up to approximately 1.5 years
  Identify systolic and diastolic readings that are outside the normal range. The number and percentage of participants who experienced significant blood pressure change from baseline will be summarized
Number of participants with change from baseline in pulse rate | Baseline up to approximately 1.5 years
  Identify pulse rate readings that are outside the normal range. The number and percentage of participants who experienced significant pulse rate change from baseline will be summarized
Number of participants with change from baseline in temperature | Baseline up to approximately 1.5 years
  Identify temperature readings that are outside the normal range. The number and percentage of participants who experienced significant temperature change from baseline will be summarized
Number of participants with change from baseline in clinical laboratory values | Baseline up to approximately 1.5 years
  Identify laboratory abnormalities from baseline will be summarized
Number of participants with change from baseline in heart rate | Baseline up to approximately 1.5 years
  Determine the effect of the drug on heart rate The number and percentage of participants who experienced heart rate changes will be summarized
Number of participants with change from baseline in QT interval | Baseline up to approximately 1.5 years
  Determine the effect of the drug on QT interval. The number and percentage of participants who experienced QT interval changes will be summarized
Number of participants with change from baseline in corrected QT interval | Baseline up to approximately 1.5 years
  Determine the effect of the drug on corrected QT interval. The number and percentage of participants who experienced corrected QT interval changes will be summarized
Number of participants with change from baseline in PR interval | Baseline up to approximately 1.5 years
  Determine the effect of the drug on PR interval. The number and percentage of participants who experienced PR interval changes will be summarized
Number of participants with change from baseline in QRS interval | Baseline up to approximately 1.5 years
  Determine the effect of the drug on QRS interval. The number and percentage of participants who experienced QRS interval changes will be summarized

SECONDARY OUTCOMES:
Number of participants with change from baseline in area under the concentration versus time curve from time zero to the last quantifiable time point (AUClast) of single ascending doses of PF-07264660 | Baseline up to approximately 1.5 years
  AUC of PF 07264660 will be calculated at selected timepoints
Number of participants with change from baseline in maximum plasma concentration (Cmax) of PF-07264660 after a single dose | Baseline up to approximately 1.5 years
  Peak concentration of PF-07264660 during selected timepoints
Number of participants with change from baseline in maximum plasma concentration (Cmax) of PF-07264660 after multiple doses | Baseline up to approximately 1.5 years
  Peak concentration of PF-07264660 during selected timepoints
Number of participants with change from baseline in time to maximum plasma concentration (Tmax) of PF-07264660 after a single dose | Baseline up to approximately 1.5 years
  Time to peak concentration of PF-07264660 during selected timepoints
Number of participants with change from baseline in time to maximum plasma concentration (Tmax) of PF-07264660 after multiple doses | Baseline up to approximately 1.5 years
  Time to peak concentration of PF-07264660 during selected timepoints
Number of participants with change from baseline in terminal elimination half-life (t½) of PF-07264660 after a single dose | Baseline up to approximately 1.5 years
  Terminal elimination half-life of PF-07264660 during selected timepoints
Number of participants with change from baseline in terminal elimination half-life (t½) of PF-07264660 after multiple doses | Baseline up to approximately 1.5 years
  Terminal elimination half-life of PF-07264660 during selected timepoints
Number of participants with change from baseline in area under the serum concentration time profile from time 0 extrapolated to infinite time (AUCinf) of single ascending doses of PF-07264660 | Baseline up to approximately 1.5 years
  AUC of PF 07264660 will be calculated at selected timepoints
Number of participants with change from baseline in area under the concentration time profile from time zero to time tau (τ), the dosing interval (AUCtau) of multiple ascending doses of PF-07264660 | Baseline up to approximately 1.5 years
  AUC of PF 07264660 will be calculated at selected timepoints
Number of participants with change from baseline in incidence and titers of anti-drug antibodies against PF-07264660 | Baseline up to approximately 1.5 years
  Number of participants with the presence of anti-PF-07264660 antibodies
Number of participants with change from baseline in incidence and titers of neutralizing antibodies against PF-07264660 | Baseline up to approximately 1.5 years
  Number of participants with the presence of anti-PF-07264660 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Collaborative Neuroscience Research, LLC, Garden Grove, California
  - Collaborative Neuroscience Research, LLC, Long Beach, California
  - Collaborative Neuroscience Research, LLC, Los Alamitos, California
  - Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Spaulding Clinical Research, West Bend, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4521001